CLINICAL TRIAL: NCT05653843
Title: MANTIS Clip Study: A Prospective, Multi-Center, All-Comer MANTIS Endoscopic Clipping Study:
Brief Title: MANTIS Endoscopic Clipping Study
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 92851066
Record Dates: First submitted 2022-06-24; First posted 2022-12-16 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Hemostasis; Perforation Colon; Feeding Tube Complication; Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Endoscopic clip placement in the gastrointestinal tract. — The placement of a mechanical endoscopic clip in the gastrointestinal tract.

SUMMARY:
This study is intended to document procedural and clinical effectiveness in consecutive cases in which at least one MANTIS clip is selected, pertaining to use of a new endoscopic clipping device MANTIS™ including but not limited to hemostasis, closure, anchoring and marking.

DETAILED DESCRIPTION:
To document clinical effectiveness and safety when used per indication within the GI tract for the purpose of:

1. Endoscopic marking
2. Hemostasis for:

   * Mucosal/sub-mucosal defects < 3 cm
   * Bleeding ulcers
   * Arteries < 2 mm
   * Polyps < 1.5 cm in diameter
   * Diverticula in the colon
   * Prophylactic clipping to reduce the risk of delayed bleeding post lesion resection
3. Anchoring to affix jejunal feeding tubes to the wall of the small bowel
4. As a supplementary method, closure of GI tract luminal perforations < 20 mm that can be treated conservatively

ELIGIBILITY:
Inclusion Criteria:

* Subject indicated for endoscopic clipping per local standard of practice.
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

* Subjects who are currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor.
* Subjects who the investigator deems at risk for study device or procedure related complications per the Instructions for Use (IFU). where commercially available or the Investigator Brochure (IB) for countries where the study device is not approved.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population will be patients usually treated for the device indication.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel von Renteln, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Jeff Mosko, MD, Principal Investigator — Unity Health Toronto
Locations (10):
- United States (4):
  - Indiana University Medical Center, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Icahn School of Medicine at Mount Sinai, New York, New York
- Canada (2):
  - St Michael's Hospital, Toronto, Onterio
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
- Shanghai Zhongshan Hospital, Shanghai, Xuhui District, China
- Prince of Wales Hospital The Chinese University of Hong Kong, Hong Kong, Shatin, Hong Kong
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India
- Showa University Koto Toyosu Hospital, Tokyo, Koto-Ku, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Renteln D, Rex DK, Pohl H, Kumta NA, Chan S, Ryou M, Nabi Z, Zhou PH, Inoue H, Peetermans JA, Rousseau MJ, Mosko JD. High Rates of Defect Closure After Resection of Large Nonpedunculated Colorectal Lesions Using a Through-The-Scope Clip With Anchor Prongs. United European Gastroenterol J. 2026 Feb;14(1):e70164. doi: 10.1002/ueg2.70164. PMID 41442239

RESULTS

PARTICIPANT FLOW:
Groups:
- MANTIS Clipping Study: Subject indicated for endoscopic clipping per local standard of practice
Period: Overall Study
Arm/Group | MANTIS Clipping Study
Started | 240
Completed | 240
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MANTIS Clipping Study
Number analyzed (Participants) | 240
Age, Continuous [Median (Standard Deviation); unit: years] | 63.4 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 217
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Hispanic or Latino data were collected for both ethnicity and race. For purposes of this Measure Hispanic or Latino were excluded from the overall count.
  Participants
    number analyzed (Participants) | 229
    American Indian or Alaska Native | 0
    Asian | 57
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 9
    White | 159
    More than one race | 0
    Unknown or Not Reported | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
Region of Enrollment [Number; unit: participants]
  Canada | 61
  Hong Kong | 23
  United States | 127
  Japan | 4
  China | 11
  India | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hemostasis of Active Bleeding
Description: Clinical success defined as hemostasis of an active bleeding assessed at the time of the index clipping procedure
Time Frame: Index Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | MANTIS Clipping Study
Number analyzed (Participants) | 240
Participants | 239

2. Primary Outcome: Number of Participants With Prophylactic Hemostasis
Description: Clinical success defined as hemostasis as a prophylactic measure to minimize risk of a delayed bleeding post lesion resection, defined as absence of a bleeding SAE up to 30 days after the index clipping procedure
Time Frame: Up to 30 Days after the index clipping procedure
Measure: Count of Participants; unit: Participants
Arm/Group | MANTIS Clipping Study
Number analyzed (Participants) | 172
Participants | 164

3. Primary Outcome: Number of Lesions With Defect Closures
Description: Clinical success defined as defect closure
Time Frame: Index Procedure
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | MANTIS Clipping Study
Number analyzed (Participants) | 240
Number analyzed (Lesions) | 249
Lesions | 4

4. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Rate of serious adverse events (SAEs) related to the MANTIS clip or the endoscopic study portion of the procedure
Time Frame: Up to 30 Days after the Endocsopic clipping procedure
Measure: Count of Participants; unit: Participants
Arm/Group | MANTIS Clipping Study
Number analyzed (Participants) | 240
Participants | 10

ADVERSE EVENTS:
Time Frame: Up to 36 days post index procedure
Arm/Group | MANTIS Clipping Study
All-Cause Mortality (participants affected / at risk) | 1/240
Serious Adverse Events (participants affected / at risk) | 14/240
Other Adverse Events (participants affected / at risk) | 0/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MANTIS Clipping Study (N=240)
Caecal perforation (Gastrointestinal disorders) | 1 (1) — Perforation: medical intervention (nothing by mouth, antibiotics. Related to Endoscopic Procedure,
Death - Worsening sepsis (Gastrointestinal disorders) | 1 (1) — Not Related to device or procedure
Aspiration (Gastrointestinal disorders) | 1 (1) — Mild related to endoscopic procedure
Diverticular bleed - site unknown (Gastrointestinal disorders) | 1 (1) — Moderate related to Endoscopic Procedure
GI Mucosal injury (Gastrointestinal disorders) | 1 (1) — Moderate related to the procedure
Intrasubmucosal leak (Gastrointestinal disorders) | 1 (1) — Moderate related to clipping procedure
Ischemia colitis (Gastrointestinal disorders) | 1 (1) — Moderate related to Endoscopic Procedure
Left lower abdominal pain (Gastrointestinal disorders) | 1 (1) — Moderate not related to clipping procedure or device
Nausea (Gastrointestinal disorders) | 1 (1) — Moderate related to Endoscopic Procedure
Ongoing lower GI bleeding (Gastrointestinal disorders) | 1 (1) — Mild bleeding related to Endoscopic Procedure
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) — Moderate related to Endoscopic Procedure
Post EMR lower GI Bleeding (Gastrointestinal disorders) | 1 (1) — Mild bleeding related to Endoscopic Procedure
Post-Polypectomy Syndrome (Gastrointestinal disorders) | 1 (1) — Moderate related to Endoscopic Procedure
Septic shock (Gastrointestinal disorders) | 1 (1) — Moderate related to the Endoscopic Procedure, Clipping Procedure, Device and the mucosotomy opening

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT05653843/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT05653843/SAP_001.pdf